CLINICAL TRIAL: NCT02402660
Title: A Phase 2 Multicenter, Double-Masked, Randomized, Placebo-Controlled Study to Investigate the Long Term Safety, Tolerability, Pharmacokinetics and Effects of ALK-001 on the Progression of Stargardt Disease
Brief Title: Phase 2 Tolerability and Effects of ALK-001 on Stargardt Disease
Acronym: TEASE
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Alkeus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK001-P1002; R01FD004098 (FDA); R01FD006016 (Other Grant/Funding Number: FDA OOPD); R01FD006316 (FDA)
Record Dates: First submitted 2015-03-09; First posted 2015-03-30 (Estimated); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Stargardt Disease; Stargardt Macular Degeneration; Stargardt Macular Dystrophy; Autosomal Recessive Stargardt Disease 1 (ABCA4-related)
MeSH Terms: conditions — Stargardt Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALK-001 (Experimental): Daily, oral administration of one capsule. See details below.
  Interventions: Drug: ALK-001
- Placebo (Placebo Comparator): Daily, oral administration of one capsule. See details below.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALK-001 — Daily, oral administration for 24 months
  Other Names: C20-D3-Retinyl Acetate; C20 Deuterated vitamin A
  Arms: ALK-001
Drug: Placebo — Daily, oral administration for 24 months
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the long term safety and tolerability of ALK-001 (C20-D3-retinyl acetate), and to explore the effects of ALK-001 on the progression of Stargardt disease in patients between the ages of 8 and 70 years old.

Funding Source - FDA OOPD

DETAILED DESCRIPTION:
This study evaluates the effects of orally-administered ALK-001 on the progression of Stargardt disease (ABCA4-related). Stargardt disease is a rare genetic disorder that leads to damage to the retina and results in legal blindness. Stargardt disease is caused by a defective ABCA4 gene, which affects the processing of vitamin A in the eye and leads to the formation of toxic vitamin A aggregates (called "vitamin A dimers") in the eye. Vitamin A dimers are thought to contribute to vision loss in Stargardt disease. ALK-001, the investigational drug, is a chemically-modified vitamin A designed as a replacement of vitamin A to prevent the formation of toxic vitamin A dimers in the eye. Trial participants will receive either ALK-001 or placebo, and follow-up visits will take place periodically for up to 24 months. There is currently no treatment for Stargardt disease.

ELIGIBILITY:
Simplified Inclusion Criteria:

* Male or female between 8 and 70 years old (inclusive), with any visual acuity
* Has a clinical diagnosis of typical autosomal recessive Stargardt macular dystrophy (STGD1)
* Has provided a genetic report indicating at least two ABCA4 disease-causing mutations. When only one ABCA4 disease-causing mutation is reported, sponsor's permission will be required.
* At least one eye (called the "primary study eye") must have at least one well-demarcated area of significantly reduced autofluorescence as imaged by fundus autofluorescence (FAF), have decreased retinal sensitivity as measured by microperimetry, or have maculopathy expected to progress over the duration of the study
* Primary study eye must have clear ocular media and adequate pupillary dilation, including no allergy to dilating eyedrops, to permit good quality retinal imaging
* Healthy as judged by investigator
* Able and willing to comply with study requirements, restrictions and instructions and is likely to complete the 24-month study
* Has signed and dated the informed consent forms (or assent where appropriate) to participate
* Female of childbearing potential has signed the informed consent about birth defects or attestation on contraception requirements

Main Exclusion Criteria:

* Has taken disallowed items (supplement containing vitamin A or beta-carotene, liver-based products, or prescription oral retinoid medications) over the past 30 days
* Is lactating, pregnant, or has a positive serum or urine pregnancy test at screening or at randomization
* Has concurrent medical condition or history, which in the opinion of the investigator, is likely to prevent compliance with the protocol and/or interfere with absorption of ALK-001 or study procedures
* Has clinically significant abnormal laboratory result(s) at screening
* Has active or historical acute or chronic liver disorder
* Has active or historical ocular disorder in the primary study eye that, in the opinion of the investigator, may confound assessment of the retina morphologically or functionally (this could include for example cataract surgery within the past 6 months, choroidal neovascularization (CNV), glaucoma, recurring uveitis, diabetic retinopathy, other retinal disease, etc.)
* Has had intraocular surgery or injections in the primary study eye within 90 days of the screening visit
* Has a clinically significant abnormal electrocardiogram (ECG), or has a corrected QT interval (QTc) that is 450 ms or greater

Ages: 8 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2015-08 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of 24 months of daily dosing of ALK-001 assessed by incidence and/or clinically significant changes of a combination of ocular and non-ocular adverse events | From baseline to 24 months

SECONDARY OUTCOMES:
Effects of ALK-001 on the progression of Stargardt disease | From baseline to 24 months
  Combination of changes in atrophic lesion size, best corrected visual acuity (BCVA), and ocular assessments.
Pharmacokinetic profile of ALK-001 derived from the concentrations of ALK-001 and metabolites in plasma | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Alkeus Site, Phoenix, Arizona
  - Alkeus Site, Los Angeles, California
  - Alkeus Site, Aurora, Colorado
  - Alkeus Site, Gainesville, Florida
  - Alkeus Site, Miami, Florida
  - Alkeus Site, Indianapolis, Indiana
  - Alkeus Site, Baltimore, Maryland
  - Alkeus Site, Grand Rapids, Michigan
  - Alkeus Site, New York, New York
  - Alkeus Site, Westbury, New York
  - Alkeus Site, Houston, Texas
  - Alkeus Site, Salt Lake City, Utah
  - Alkeus Site, Silverdale, Washington
  - Alkeus Site, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ma L, Kaufman Y, Zhang J, Washington I. C20-D3-vitamin A slows lipofuscin accumulation and electrophysiological retinal degeneration in a mouse model of Stargardt disease. J Biol Chem. 2011 Mar 11;286(10):7966-7974. doi: 10.1074/jbc.M110.178657. Epub 2010 Dec 14. PMID 21156790
- [Background] Kaufman Y, Ma L, Washington I. Deuterium enrichment of vitamin A at the C20 position slows the formation of detrimental vitamin A dimers in wild-type rodents. J Biol Chem. 2011 Mar 11;286(10):7958-7965. doi: 10.1074/jbc.M110.178640. Epub 2010 Nov 12. PMID 21075840
- [Background] Mihai DM, Jiang H, Blaner WS, Romanov A, Washington I. The retina rapidly incorporates ingested C20-D(3)-vitamin A in a swine model. Mol Vis. 2013 Jul 25;19:1677-83. Print 2013. PMID 23914132
- [Background] Charbel Issa P, Barnard AR, Herrmann P, Washington I, MacLaren RE. Rescue of the Stargardt phenotype in Abca4 knockout mice through inhibition of vitamin A dimerization. Proc Natl Acad Sci U S A. 2015 Jul 7;112(27):8415-20. doi: 10.1073/pnas.1506960112. Epub 2015 Jun 23. PMID 26106163
- [Background] Saad L, Washington I. Can Vitamin A be Improved to Prevent Blindness due to Age-Related Macular Degeneration, Stargardt Disease and Other Retinal Dystrophies? Adv Exp Med Biol. 2016;854:355-61. doi: 10.1007/978-3-319-17121-0_47. PMID 26427432
- [Background] Zhang D, Robinson K, Washington I. C20D3-Vitamin A Prevents Retinal Pigment Epithelium Atrophic Changes in a Mouse Model. Transl Vis Sci Technol. 2021 Dec 1;10(14):8. doi: 10.1167/tvst.10.14.8. PMID 34878528
- [Background] Zhang D, Robinson K, Saad L, Washington I. Vitamin A cycle byproducts impede dark adaptation. J Biol Chem. 2021 Sep;297(3):101074. doi: 10.1016/j.jbc.2021.101074. Epub 2021 Aug 12. PMID 34391781
- See also: Please leave your name if you would like to be contacted to discuss this trial — http://www.alkeuspharma.com/contact-us/